CLINICAL TRIAL: NCT06966258
Title: Inspire HER: Inspiring the Heart and Emotions for Radical Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other); Ohio State University (Other); Tuskegee University (Other)
Responsible Party: Principal Investigator, Timiya Nolan, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300014631; 25SFRNPCKMS1468507 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular-kidney-metabolic Syndrome; Cardiovascular Diseases; Hypertension; Diabetes; Hyperlipidemia; Kidney Disease; Obesity; Smoking
Keywords: Cardiovascular Risk; Lifestyle intervention
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Hyperlipidemias; Kidney Diseases; Obesity; Smoking

STUDY DESIGN:
Intervention Model Description: Randomized, wait-list controlled trial
Who Masked: Outcomes Assessor
Masking Description: The statistical analyst is blinded to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspire HER Intervention (Experimental): Those in the Inspire Her intervention arm will receive the 24-week intervention.
  Interventions: Behavioral: Inspire HER Intervention
- Wait-list Control (No Intervention): Those in the wait-list control arm will receive usual care.

INTERVENTIONS:
Behavioral: Inspire HER Intervention — The Black Impact intervention is an academic-community-government partnership adapted from the Diabetes Prevention Program and American Heart Association Check, Change, Control programs based on stakeholder feedback and to afford incorporation of additional evidence-based strategies for influencing target outcomes. The intervention is a 24-week community-based lifestyle intervention to improve cardiovascular health among Black men. Each participant will be assigned to a group with >5 participants based on participant proximity to a central community meeting location. Each team will be guided weekly by a health coach who delivers content and coaching around the lifestyle intervention modeled on the diabetes prevention program and check, change, control blood pressure program, a community health worker who helps to address social needs and connects participants to primary care services, and a trainer who leads physical activity. Teams meet for 90 minutes per week.
  Arms: Inspire HER Intervention

SUMMARY:
Poor heart health puts Black women at risk for a shorter life with more illness than people of any other non-indigenous racial group. We will refine and conduct a randomized, wait-list controlled trial of Inspire HER (a heart health lifestyle intervention for Black women that provides health education, physical activity, and social resources). We will also compare Inspire HER and Black Impact (a heart health intervention for Black men) data to study how women and men respond differently to stress. This trial aligns with American Heart Association's pledge to address heart health equity through new interventions that consider the person and the circumstances with which they live.

DETAILED DESCRIPTION:
Poor heart health puts Black women at risk for a shorter life with more illness than people of any other non-indigenous racial group. Yet, few studies have focused on improving heart health in Black women. Our team built and studied a 24-week program called Black Impact for Black men with less than ideal heart health. Black Impact provides 45 minutes of exercise and 45 minutes of healthy diet education and connects Black men with a health coach, fitness trainer, and community health worker. In the first study of Black Impact, Black men (n=74) had improved heart health equal to a 19% lower risk of death from heart disease. These men also reported less stress, improvement in being able to control their health, and fewer unmet social needs. Now, a study of Black Impact in 340 Black men is ongoing to understand how Black Impact works with respect to stress and heart health. Black women have reported a need for a similar heart health program. Based on feedback from Black women (n=56), we adapted Black Impact for Black women (Inspire HER). Thus, we propose to refine the Inspire HER program for Black women. Then, we will do a clinical trial of Inspire HER compared to routine living (usual care) in Black women with elevated heart health risk. We will find out if the Inspire HER program reduces heart health risk more than usual care. We will also assess how the Inspire HER program "gets under the skin" to affect the body's response to stress. Lastly, we will compare the response to stress between women of Inspire HER and men of Black Impact. Importantly, we expect this study will show promising improvements in heart health and risk. This Inspire HER trial will lay the foundation for larger future studies. Inspire HER, comparing data from Black Impact, may also help us understand how women and men in heart health programs respond differently to stress. This trial aligns with American Heart Association's pledge to address heart health equity through new interventions that consider the person and the circumstances with which they live.

ELIGIBILITY:
Inclusion Criteria:

* Black women (self-report)
* Adult ages 30-79 years
* Stage 2 or greater Cardiovascular-Kidney-Metabolic Syndrome
* English speaking
* Lives in Metropolitan Birmingham, AL area.

Exclusion Criteria:

- Healthcare provider-imposed physical activity limitations.

Ages: 30 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Preliminary Effect on PREVENT Score) | 24 weeks
  The primary outcome for the randomized controlled trial is change in cardiovascular risk as defined by PREVENT Score (a 10-year risk estimator of cardiovascular events for individuals 30-79 years of age; measure utilizes sex, age, cholesterol blood pressure, body mass index, glomerular filtration rate, diabetes, smoking status, anti-hypertensive medication, lipid-lowering medication, urine creatinine, hemoglobin A1C, and social deprivation index). PREVENT score ranges from low (<5%) to high (>20%) risk with low risk being better. Linear mixed effects models with random intercepts will evaluate the change from baseline to 24 weeks in primary (PREVENT score). These models will assess differences between waitlist control and intervention participants using an interaction between time and treatment indicator. We will also evaluate qualitative exit (focus group) survey data to understand perceived effect.
Feasibility (Demand or Use of Intervention) | 24 weeks
  Demand will be assessed by percent recruited of number contacted, participant self-rating of participation, percent using information at home. These data will be obtained from study records and exit survey (focus group) responses.
Feasibility (Acceptability or Participant Reaction to Intervention) | 24 weeks
  Acceptability will be assessed by participant satisfaction with the intervention and participant attendance, perceptions of usefulness, and plans/real change of behavior to apply health promotion strategies. These data will be obtained by study records and exit (focus group) surveys.
Feasibility (Implementation or Intervention FIdelity) | 24 weeks
  Implementation will be assessed using the Inspire HER curriculum and participant opinions of how the intervention was administered. These data will be obtained via study records and exit (focus group) surveys.
Feasibility (Practicality or Efficiency of Resource Allocation) | 24 weeks
  Practicality will be assessed using intervention cost per participant and identifying any revenue/savings. These data will be obtained by evaluating grant budgetary documentation.

SECONDARY OUTCOMES:
Dose-Response on Preliminary Effect | 24 weeks
  Dose-response will be assessed by studying the relationship between intervention engagement (i.e. attendance) and the primary study outcome (change in PREVENT score). These data will be obtained using study records and PREVENT score evaluation as identified in the primary outcome.
Change in Conserved Transcriptional Response to Adversity | 24 weeks
  Evaluation of change in conserved transcriptional response to adversity (CTRA) will be measured via collection of blood and measuring leukocyte gene expression to determine the CTRA at baseline, 12 and 24 weeks. For the CTRA score, background subtraction and normalization of raw data, and operationalize inflammatory and antiviral gene activity will be performed. CTRA change will be calculated using between-subject differences using a linear mixed-effects to evaluate changes from baseline. The model will contain data from baseline (0 weeks), during-intervention (12 weeks), and post-intervention (24-weeks). These models will assess differences between waitlist control and intervention participants using an interaction between time and treatment indicator. Residual plots will examine model assumptions and model fit, with transformation of the outcomes used as needed to satisfy modelling assumptions and achieve appropriate model fit.
Change in 12,13-diHOME Expression and Associations with Biomarkers | 24 weeks
  Evaluation of change in 12,13-diHOME expression will be measured via collection of blood and measuring leukocyte gene expression to determine the expression at baseline, 12 and 24 weeks. For the expression score, background subtraction and normalization of raw data, and operationalize inflammatory and antiviral gene activity will be performed. The expression change will be calculated using between-subject differences using a linear mixed-effects to evaluate changes from baseline. The model will contain data from baseline (0 weeks), during-intervention (12 weeks), and post-intervention (24-weeks). These models will assess differences between waitlist control and intervention participants using an interaction between time and treatment indicator. Residual plots will examine model assumptions and model fit, with transformation of the outcomes used as needed to satisfy modelling assumptions and achieve appropriate model fit.
Mechanistic transcriptomic stress and inflammatory response to Inspire HER in Black women as compared to Black men in Black Impact: | 24 weeks
  Heterogeneity of treatment differences between women enrolled in the Inspire HER study and men enrolled in the Black Impact 2.0 study (NCT: NCT06055036) will be examined visually using lattice graphical displays. ComBat will evaluate and address potential batch effects in CTRA (as described in the secondary outcome above) data between the two studies. Linear mixed models will estimate potential heterogeneity in response by sex via inclusion of sex*treatment interaction terms.

CONTACTS AND LOCATIONS:
Overall Officials: Timiya S Nolan, PhD, Principal Investigator — University to Alabama at Birmingha
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 3/31/2025; available without end date
Access Criteria: Inspire HER will generate primary qualitative and quantitative data. Qualitative data will be derived from focus group interviews with participants and partners of the Inspire HER intervention. To facilitate data interpretation, documentation files (txt files) such as a data dictionary, interview and survey questionnaires, informed consent script and study protocol will be made publicly available via Dryad. Quantitative data will be derived from participants' survey responses about cardiometabolic and social health. We will produce data management and analytic files (CSV files) that will be posted on GitHub.
  Because of the sensitive nature of community-based research, policies and guidelines will require having a faculty member with expertise in health equity research, IRB approval, and a community partner to help interpret findings and create/enact a dissemination plan.

REFERENCES:
- [Background] Joseph JJ, Nolan TS, Williams A, McKoy A, Zhao S, Aboagye-Mensah E, Kluwe B, Odei JB, Brock G, Lavender D, Gregory J, Gray DM 2nd. Improving cardiovascular health in black men through a 24-week community-based team lifestyle change intervention: The black impact pilot study. Am J Prev Cardiol. 2022 Jan 13;9:100315. doi: 10.1016/j.ajpc.2022.100315. eCollection 2022 Mar. PMID 35146467